CLINICAL TRIAL: NCT07083804
Title: Feasibility Study to Diagnose Helicobacter Pylori In The Paediatric Population Using Non-Invasive Fecal Analysis: the HEPYCA Study
Brief Title: Feasibility Study to Diagnose Helicobacter Pylori in the Paediatric Population Using Non-invasive Fecal Analysis
Acronym: HEPYCA
Status: Recruiting | Type: Observational
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-A02366-41
Record Dates: First submitted 2025-07-11; First posted 2025-07-24 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-07

CONDITIONS: HELICOBACTER PYLORI INFECTIONS
Keywords: Pediatrics; Gastroenterology; Microbiology; Infectious disease; Helicobacter pylori
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Days
Biospecimen Retention: Samples Without DNA — Gastric biopsy and stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric patients: Pediatric patients consulted/hospitalized for sampling for the presence or absence of Helicobacter pylori.
  Interventions: Diagnostic Test: Gastric biopsies; Diagnostic Test: Stool sampling

INTERVENTIONS:
Diagnostic Test: Gastric biopsies — After obtaining informed consent, patients receive routine endoscopic procedures with an additional biopsy taken for research purposes.
  Invasive screening method used in routine care.
Diagnostic Test: Stool sampling — Stool samples are taken and sent within 10 days of the endoscopy. Self-collected stool samples are analyzed using antigen testing and molecular techniques to detect H. pylori and associated resistance mutations.
  Experimental diagnosis.

SUMMARY:
Helicobacter pylori infection is a widespread bacterial disease affecting nearly half of the world's population. In children, the infection displays distinct features versus adults, with lower prevalence, variable symptoms, and differing endoscopic and histological appearances.

Typically acquired in early childhood, its transmission is closely linked to socio-economic disadvantage and overcrowding. Although most infected children are asymptomatic, some develop epigastric pain, dyspepsia, weight loss, or other gastrointestinal disturbances. Chronic infection may eventually lead to mucosal atrophy and intestinal metaplasia, increasing the risk of gastric cancer later in life. Given the limitations and risks of invasive diagnostic methods-especially endoscopy under general anesthesia-there is a critical need for reliable, non-invasive tests. Recent adult studies indicate that stool-based PCR is a promising alternative for both detecting H. pylori and identifying clarithromycin resistance.

The primary objectives of this study are to evaluate the intrinsic diagnostic performance of high-resolution melt PCR (HP PCR) in stools, and to compare these results with those obtained from a conventional work-up, such as gastric biopsies, in a paediatric population. In accordance with prevailing rationality, the principal outcome of this study will be an evaluation of the intrinsic diagnostic capabilities of the proposed method. This will be accomplished by conducting a comparison of the sensitivity and specificity of the PCR test in stools with those of gastric biopsies (reference test).

ELIGIBILITY:
Inclusion Criteria:

* Age < or = 16 years ;
* Any indication for gastroscopy in children requiring gastric biopsies: gastro-esophageal reflux resistant to proton pump inhibitors (PPIs) or recurrent on discontinuation of PPIs, hematemesis, refractory anemia or unexplained inflammatory syndrome, recurrent vomiting, dysphagia, endoscopic assessment of chronic inflammatory bowel disease with search for H. pylori superinfection ;
* Patients benefiting from a Social Security scheme or benefiting from one via a third part;
* Holders of parental authority who have given their informed consent to participate in the study and child participants of understanding age who have given their assent.

Non-inclusion Criteria:

* Antibiotic treatment less than 4 weeks
* PPIs treatment less than 2 weeks
* Contraindication to endoscopic procedure or biopsy.

Exclusion Criteria:

* Antibiotic therapy prior to stool collection (between inclusion and stool collection, which may be 10 days later)
* Failure to send/receive stool sample
* Biopsy not performed at endoscopy

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children requiring gastric biopsies for H. pylori detection
Sampling Method: Non-Probability Sample
Enrollment: 188 (Estimated)
Dates: Start 2025-10-07 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Evaluate the diagnostic performance of H. pylori PCR in stools | 10 days
  Diagnostic capabilities will be assessed by the error rate (false positives and negatives) of the stool PCR test, compared with the results of PCR biopsy (reference test).

SECONDARY OUTCOMES:
Evaluate the intrinsic diagnostic performance (Se, Sp) of H. pylori PCR in stools | 10 days
  Intrinsic diagnostic capabilities will be assessed by comparing the sensitivity and specificity of the stool PCR test with the results of gastric biopsies (reference test).
Evaluate the extrinsic diagnostic performance (PPV, NPV) of H. pylori PCR in stools | 10 days
  Extrinsic diagnostic capabilities will be assessed by comparing the positive and negative predictive values of the stool PCR test with the results of gastric biopsies (reference test).
Evaluate the intrinsic diagnostic performance (Se, Sp) of clarithromycin-resistant H. pylori PCR in stools | 10 days
  Intrinsic diagnostic capabilities will be assessed by comparing the sensitivity, specificity and positive and negative predictive values of the clarithromycin-resistant H. pylori PCR test in stools with those of gastric biopsies (reference test).
Evaluate the extrinsic diagnostic performance (PPV, NPV) of clarithromycin-resistant H. pylori PCR in stools | 10 days
  Extrinsic diagnostic capabilities will be assessed by comparing the sensitivity and specificity, as well as the positive and negative predictive values, of the clarithromycin-resistant H. pylori PCR test in stools with the results of gastric biopsies (reference test).
Evaluate the intrinsic and extrinsic diagnostic performance of H. pylori PCR and H. pylori antigen in stools | 10 days
  Intrinsic and extrinsic diagnostic capabilities will be assessed by comparing the sensitivity and specificity and positive and negative predictive values of the stool antigen test with the results of gastric biopsies (reference test).
Evaluate the intrinsic diagnostic performance (Se, Sp) of H. pylori PCR in stools | 10 days
  Intrinsic diagnostic capabilities will be assessed by the sensitivity and specificity and positive and negative predictive values of the stool PCR test, and compared with stool antigen results.
Evaluate the extrinsic diagnostic performance (PPV, NPV) of H. pylori PCR in stool | 10 days
  Extrinsic diagnostic capabilities will be assessed by the sensitivity and specificity and positive and negative predictive values of the stool PCR test, and compared with stool antigen results.
Evaluate the adherence of a stool self-sampling for H. pylori | 10 days
  Adherence to stool sampling will be assessed by the number of stool samples received in the population analyzed out of the number of patients included
Analyze resistance profiles to the various antibiotics used in Helicobacter pylori eradication therapy | 10 days
  Analyze resistance profiles to the various antibiotics used in Helicobacter pylori eradication therapy in relation to biological test results (PCR in biopsy and stool, stool antigens) and clinical presentation. Resistance profiles will be expressed in micrograms per mL and interpreted in accordance with the current guidelines of the Antibiogram Committee of the French Microbiology Society.

CONTACTS AND LOCATIONS:
Locations (1):
- Poitiers University Hospital, Poitiers, France

IPD SHARING:
Plan to Share IPD: No